CLINICAL TRIAL: NCT02143336
Title: Prospective and Comparative Pilot Study Between Subcuticular Continuous Suture Versus Skin Staples to Reduce Surgical Site Infections in Colorectal Surgery Patients.
Brief Title: Subcuticular Continuous Suture Versus Skin Staples to Reduce Surgical Site Infections in Colorectal Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Surgical Infection Society Europe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HULP-3961
Record Dates: First submitted 2014-05-17; First posted 2014-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Surgical Wound Infections; Colorectal Surgery
Keywords: Surgical site infections; Skin closure techniques; Colorectal surgery
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcuticular suture (Experimental): Subcuticular suture (absorbable) for skin closure
  Interventions: Procedure: subcuticular suture
- Skin staples (Active Comparator): Standard skin staples for wound closure
  Interventions: Procedure: Skin staples

INTERVENTIONS:
Procedure: subcuticular suture
  Other Names: undyed Monocryl 4-0 (Ethicon)
  Arms: Subcuticular suture
Procedure: Skin staples
  Arms: Skin staples

SUMMARY:
A comparison of skin closure techniques (standard skin closure with staples versus a continuous (subcuticular) absorbable suture), to determine if this changes the rate of post operative wound infections in elective colorectal surgery patients.

DETAILED DESCRIPTION:
In colorectal surgery, there has been a growing interest in the study of Surgical Site Infections (SSI), with an outstanding variability of reported incidence, ranging from 3% up to 30% depending on the series. Although general risk factors for infection have been identified, there is still a need to identify specific risk factors for colorectal surgery patients, to try to reduce these numbers. The technique and materials used for wound closure have been considered as interesting variables for study.

Main question of our study: is subcuticular (reabsorbable, continuous) suture better than skin staples for reducing wound SSIs in colorectal surgery? The study is sponsored by the Surgical Infection Society Europe, and was awarded the SIS-E Fellowship for young investigators (2013)

ELIGIBILITY:
Inclusion Criteria:

* Adults (age >18), both genders.
* Elective colorectal surgery interventions
* Open surgery incisions and laparoscopic extraction incisions
* Incisions >5cm, any location
* Intervention performed by a specialist colorectal surgeon
* Patient suitable for surgery in preoperative assessment
* Informed consent

Exclusion Criteria:

* Emergency colorectal surgery
* Scheduled multiple surgical procedures
* Unsuitable preoperative assessment
* Other infections present/being treated.
* Incorrect application of standard surgical infection prevention measures (antibiotic prophylaxis, antibiotic treatment prior to surgery, intraoperative heat/O2/glycemic control,etc.)
* Inability to understand the study/sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
incidence of surgical site infection | 30 days, as by CDC definition
  The primary endpoint is the incidence of wound infection, measured from the moment of surgery up to 30 days postoperatively.

SECONDARY OUTCOMES:
prolongation of hospitalization | 30 days
  Length of hospital stay, and if it is prolonged as a consequence of infection

CONTACTS AND LOCATIONS:
Overall Officials: Ines Rubio-Perez, MD, Principal Investigator — Hospital Universitario La Paz
Locations (2):
- Spain (2):
  - Hospital Fundacion Jimenez Diaz, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid

REFERENCES:
- See also: Surgical Infection Society Europe, main webpage — http://www.sis-e.org/